CLINICAL TRIAL: NCT03421899
Title: Systems Medicine of Mitochondrial and Biochemical Parkinson's Disease and Other Related Movement Disorders
Brief Title: A Study Into the Underlying Biochemical Pathways Involved in Parkinson's Disease, Such as Mitochondrial (Cellular "Powerhouse") Dysfunction
Acronym: SysMedPD
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: European Commission (Other); University of Luxembourg (Other); University of Luebeck (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0126
Record Dates: First submitted 2017-11-23; First posted 2018-02-05 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Parkinsonism
Keywords: Mitochondria; Mitochondrial dysfunction; Parkin; PINK1
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (DNA and RNA), plasma, serum, urine, cerebrospinal fluid (CSF), skin (as fibroblast cell lines) and fat (as adipose stem cell lines)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Genetic Parkinson's group: Those participants with Parkinson's disease and a genetic mutation known to cause or increase risk of Parkinson's disease (e.g. Parkin, PINK1, GBA or LRRK2)
- Idiopathic Parkinson's group: Those participants with Parkinson's disease but without a known genetic mutation known to cause or increase risk of Parkinson's disease
- Healthy control group: Those participants unaffected by Parkinson's disease

SUMMARY:
Parkinson's disease (PD) is a progressive neurological disorder that is increasingly common with age, with the incidence rising from approximately 4 people per 10,000 in their forties to 2 in 100 over the age of eighty.

Our understanding of the causes of PD has rapidly developed in the past two decades, but this has not yet translated into any clinically established neuroprotective treatment that slows disease progression. There is a growing consensus that the failure of previous efforts is mainly due to the causative diversity of PD i.e. that PD may have many different causes. For example, it is known that variants in mitochondrial (cellular power house) genes can cause specific forms of PD and this may be relevant to other forms of PD.

The aim of this study is to attempt to group PD patients based on markers of biochemical dysfunction (e.g. into groups of patients that do and those who do not have evidence of mitochondrial dysfunction) to aid in the development of new candidate neuro-protective compounds.

The investigators hope by grouping people with Parkinson's into those with and without impaired mitochondrial function the investigators will be better able to develop more targeted treatments aimed at protecting further loss of brain cells that occurs in Parkinson's disease.

To achieve this the investigators will study people, in two study sites in London, with both genetic forms of PD and those with idiopathic PD (i.e. those where there is not a known genetic variant causing PD), as well as a healthy control group. All groups will undergo standardised clinical assessment to collect information on several aspects of their condition (e.g. disease severity, memory problems and sleep problems).

Participants will be asked to provide blood, urine and optionally cerebrospinal fluid & skin samples from which various biochemical assays and genetic analysis will be performed in attempt to group participants based on the results of these tests. The study is funded for 3 years with participants being asked to attend for up to 3 study visits each over this time period.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurological disorder that is increasingly prevalent with age, with the incidence rising from approximately 4 people per 10,000 in their forties to 2 in 100 over the age of eighty. Besides motor symptoms, such as tremor, rigidity, bradykinesia, and postural instability, PD patients often experience a variety of non-motor symptoms, such as fatigue, depression, sleep disturbance, and dementia.

Although symptomatic treatments exist to partially compensate for motor dysfunction, no neuroprotective treatment has yet been established to slow PD progression, which inevitably renders patients incapable of living independently. Compared to age- and sex-matched controls, PD patients are about 5 times more likely to require nursing home care and this care costs about 5 times more than average nursing home care. This, combined with the European demographic shift toward an increasingly larger fraction of aged individuals, creates a social and economic challenge to develop new medications to slow the progression of PD.

Our understanding of the aetiopathogenesis of PD has rapidly developed in the past two decades, but this has not yet translated into any clinically established neuroprotective treatment that slows disease progression. There is a growing consensus that the failure of previous efforts is mainly due to the aetiopathogenic diversity of PD and the estrangement of existing preclinical models from clinical PD. For example, it is known that mutations in mitochondrial genes can cause monogenic PD and biochemical evidence indicates that in a proportion of cases, idiopathic PD is associated with detectable mitochondrial dysfunction.

Therefore, the investigators focus is on monogenic forms of PD that involve mitochondrial abnormalities as a primary (e.g., Parkin, PINK1), or secondary (e.g., LRRK2, GBA1) phenomenon, in order to extrapolate to idiopathic PD (IPD) patients with and without mitochondrial dysfunction (Mito-IPD and Amito-IPD, respectively). Biochemical pathways focusing on, but not restricted to mitochondrial function, will be assessed using a variety of techniques including biochemical assays on blood, urine, CSF and tissue samples. The investigators will explore both the relevance and measurement of specific biochemical pathways in Parkinson's and related disorders

The main overall objective is to stratify PD patients based on dysfunction in biochemical pathways related to PD. This will aid in developing new candidate neuroprotection compounds to slow the progression of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PD, or a related condition (e.g. Parkinson's plus, dystonia, tremor) or healthy control participant
2. Age 18 years or over

Exclusion Criteria:

1. Lack of capacity to consent to participate in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of people with PD (those with and without know genetic mutations associated with PD) as well as an age matched control population.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Definition of a reproducible biochemical method of grouping people with Parkinson's based on defined biochemical dysfunction | 3 years
  The study will primarily aim to stratify patients by the degree of mitochondrial dysfunction detected by a battery of functional assays.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Schapira, Principal Investigator — UCL Institute of Neurology; Huw Morris, Principal Investigator — UCL Institute of Neurology
Locations (1):
- UCL Institute of Neurology, Department of Clinical Neurosciences, Upper 3rd Floor, Royal Free Hospital, Rowland Hill Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT03421899/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT03421899/SAP_001.pdf
  • Informed Consent Form (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT03421899/ICF_002.pdf